CLINICAL TRIAL: NCT01723748
Title: Somatostatin Analogue Treatment of Acromegaly: Molecular Aspects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-491-12; 35197 (Other: VEK)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2014-12

CONDITIONS: Acromegaly; Metabolic Diseases
Keywords: Acromegaly; Somatostatin treatment; metabolic effect
MeSH Terms: conditions — Acromegaly; Metabolic Diseases | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery treated (Active Comparator): 10 patients with well-controlled acromegaly for at least 6 months after surgery alone.
  Stimulated with genotropin
  Interventions: Drug: genotropin
- SA treated (Active Comparator): 10 patients with well-controlled acromegaly for at least 6 months after SA treatment Stimulated with genotropin
  Interventions: Drug: genotropin

INTERVENTIONS:
Drug: genotropin — iii) intravenous exogenous bolus of GH (0.5 mg) followed by muscle and fat biopsies.
  Other Names: growth hormone

SUMMARY:
The treatment with SA still leaves some questions unanswered. Firstly, SA treatment often results in a concomitant suppression of the insulin secretion, which might lead to clinically significant glucose intolerance. Secondly, the traditional evaluation of disease activity by measuring circulating levels of GH and total IGF-I is not reliable enough

Hypotheses: Treatment of acromegaly with SA versus surgery alone is associated with:

* Glucose intolerance despite normalized insulin sensitivity
* Modified peripheral GH activity in peripheral target organs assessed on molecular endpoints

DETAILED DESCRIPTION:
Acromegaly is a rare disease usually caused by a benign growth hormone (GH) producing pituitary adenoma. In case of inadequate disease control, the condition is associated with significant morbidity and approximately a doubling of mortality compared to the background population. Medical treatment with somatostatin analogues (SA) has been employed for about 20 years and is a well-established treatment in cases where surgery is impossible or inadequate. The treatment with SA still leaves some questions unanswered. Firstly, SA treatment often results in a concomitant suppression of the insulin secretion, which might lead to clinically significant glucose intolerance. Secondly, the traditional evaluation of disease activity by measuring circulating levels of GH and total IGF-I is not reliable enough

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* treated acromegaly
* considered suitable

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Metabolism - including GH, IGF-I, FFA, glc and insulin. Concentration and AUC (area under the curve) | 3 years
  GH (ug/l), IGF-I (ug/l), FFA (mmol/l) , glc (mmol/l) and insulin (pmol/l)

SECONDARY OUTCOMES:
concentration of serum and interstitial GH, bioactive IGF-I as well as total IGF-I | 3 years
  GH (ug/l), IGF-l (ug/l), bioactive IGF-l (ug/l)

OTHER OUTCOMES:
GH, and insulin signal transduction in muscle and fat biopsies and regulation of lipolysis. | 3 years
  By western blot technique protien levels of (arbitrary densitomety units) AKT, pAKT threonin, pAKT serine, STAT5, pSTAT5, PTEN, p85alpha, mTOR, pmTOR.
  By PCR technique (relative nRNA expression) mRNA levels of IGF-1, SOCS1, SOCS2, SOCS3, CISH, PTEN, Pik3r
patient characterization | 3 years
  sex (M/F), age (year), disease duration (years), BMI (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Joergensen, professor, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No